CLINICAL TRIAL: NCT02636933
Title: Longitudinal Observational Study in Prematurely Born Preschool Children: Assessment of Lung Function Parameters (PRE-AR) (PREMATURELY BORN CHILDREN- ASTHMA AND ALLERGIC RHINITIS )
Brief Title: Longitudinal Observational Study in Prematurely Born Preschool Children: Assessment of Lung Function Parameters
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Stefania La Grutta, MD (Other)
Responsible Party: Sponsor-Investigator, Stefania La Grutta, MD, Stefania La Grutta, MD. Senior Researcher. Coordinator of Pediatric Allergy and Asthma Research Group. Institute of Biomedicine and Molecular Immunology, IBIM, National Research Council of Palermo, Italy., Istituto per la Ricerca e l'Innovazione Biomedica
Organization: Istituto per la Ricerca e l'Innovazione Biomedica (Other)
Other Study IDs: 9/2014
Record Dates: First submitted 2015-10-02; First posted 2015-12-22 (Estimated); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Asthma; Allergic Rhinitis
Keywords: Asthma; Allergic Rhinitis; Children; Atopy
MeSH Terms: conditions — Asthma; Rhinitis, Allergic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 59 prematurely born children: Lung function assessment of 59 prematurely born children (of both sex and 3-5 years old) attending as outpatient clinic of Pediatric Allergology & Pulmonology (PAP) of Respiratory Disease Research Center (RDRC) within the Institute of Biomedicine and Molecular Immunology (IBIM) of the National Research Council (CNR) of Palermo (RDRC-IBIM CNR)
  Interventions: Other: Lung Function Assessment
- 93 full-term born children: Lung function assessment of a Control group of full-term born children (N=93), recruited by a collaborative Pediatricians network within the Institute of Biomedicine and Molecular Immunology (IBIM) of the National Research Council (CNR) of Palermo (RDRC-IBIM CNR), Italy.
  Interventions: Other: Lung Function Assessment

INTERVENTIONS:
Other: Lung Function Assessment — Lung Function Assessment

SUMMARY:
The PRE-AR project is a longitudinal observational study. The primary objective is the assessment of lung function parameters in late preterm preschool children.

DETAILED DESCRIPTION:
The PRE-AR project is a longitudinal observational study. The primary objective is the assessment of lung function parameters in late preterm preschool children.

Pulmonary function tests will be performed.

ELIGIBILITY:
Case group

Inclusion Criteria:

* Premature birth < 37 weeks
* 5 years old ≤ Age ≥ 3 years old

Control group

Inclusion Criteria:

* Full-term birth
* 5 years old ≤ Age ≥ 3 years old

Exclusion Criteria of both groups:

* Pulmonary bronchodysplasia (BDP)
* Acute respiratory infection
* Immunological and metabolic system disease
* Malformation of upper respiratory tract
* Topical or systemic therapies, with antibiotics, antihistaminics and corticosteroids, in the previous 30 days
* Patients with neurological pathologies
* Patients that are not able to perform the lung function tests

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: A study population of 59 prematurely born children (of both sex and 3-5 years old) attending as outpatient clinic of Pediatric Allergology & Pulmonology (PAP) of Respiratory Disease Research Center (RDRC) within the Institute of Biomedicine and Molecular Immunology (IBIM) of the National Research Council (CNR) of Palermo (RDRC-IBIM CNR).
  A Control group of full-term born children (N=93), recruited by a collaborative Pediatricians network within the Institute of Biomedicine and Molecular Immunology (IBIM) of the National Research Council (CNR) of Palermo (RDRC-IBIM CNR), Italy.
  The subjects will be paired up according to the sex and to the age, with a ratio 1:1.
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2015-03; Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Forced oscillation technique | Baseline, 24 months, and 48 months
  Longitudinal assessment of forced oscillation technique (FOT)
Spirometry | Baseline, 24 months, and 48 months
  Longitudinal assessment of spirometry
Interrupter resistance | Baseline, 24 months, and 48 months
  Longitudinal assessment of interrupter resistance (RINT)

SECONDARY OUTCOMES:
Nasal nitric oxide | Baseline, 24 months, and 48 months
  Longitudinal assessment of nasal nitric oxide (nNO)
Atopy | Baseline
  Positivity to at least one aeroallergen
Nasal brushing | Baseline
  Assessment of alterations and inflammatory changes in the nasal mucosa
Saliva sample | 24 months, and 48 months
  Phenotypic characterization through the collection of saliva samples
Urine analysis | Baseline, 24 months, and 48 months
  Endotypic characterization through urine proteomic analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Biomedicine and Molecular Immunology, IBIM, Palermo, Italy

IPD SHARING:
Plan to Share IPD: Yes
The IPD collected will be available on december 2020.
  The following participant data will be shared:
  * Pulmonary function tests
  * Demographic characteristics
  All IPD will be obtained from statistical analysis on the dedicated database in which all data are stored.